CLINICAL TRIAL: NCT04362956
Title: Clinical and Immunologic Impact of SARS-CoV-2 in Hospitalized Pregnant Women and Neonates in Argentina
Brief Title: Clinical and Immunologic Impact of Perinatal SARS-CoV-2 (COVID-19) Infection
Status: Completed | Type: Observational
Sponsor: Fundacion Infant (Other)
Responsible Party: Sponsor
Other Study IDs: Perinatal COVID-19
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Pregnancy Related; Neonatal Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal aspirates Maternal serum Umbilical Cord serum Human milk
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a multi-center prospective study that aims to investigate the clinical and immunologic impact of SARS-CoV-2 infection in pregnant women and neonates. The goal is to recruit 200 SARS-CoV-2 infected pregnant women starting at 24 weeks of gestation in a neonatal network of 45.000 birth a year. Clinical data will be collected from women and neonates. Upper airways samples will be obtained from both for bio-markers investigation. Finally, maternal and umbilical cord serum and human milk will be obtained for antibody assessment.

DETAILED DESCRIPTION:
COVID-19, the disease caused by the novel coronavirus SARS-CoV-2, has led to an unprecedented global pandemic affecting persons of all ages. Pregnant women are in a physiologic immunosuppressed situation and have a greater risk and severity of respiratory infection. However, considerable uncertainty exists regarding the potential for vertical transmission (prenatal/congenital or perinatal) of SARS-CoV-2 from infected pregnant women to their newborns and its potential clinical consequences.

This study attempts to provide evidence-based guidelines for managing antenatal, intrapartum, and neonatal care around COVID-19 require an understanding of whether the virus can be transmitted transplacentally; a determination of which maternal body fluids may be infectious; trasnplacental and human milk antibody transfer and data of adequate statistical power that describe which maternal, intrapartum, and neonatal factors influence perinatal transmission.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women hospitalized presenting with:

  1. Fever with one or more respiratory symptoms (cough, odinophagia, respiratory difficulty)
  2. Diagnoses of pneumonia with no other explainable cause.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Elegible patients will be all pregnant women of 9 large maternity hospitals in Argentina.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Vertical transmission | 96 hours from birth
  Presence of IgM in Umbilical Cord or presence of virus in human milk with infected neonate
Neonatal protection due to maternal antibodies | 24 weeks of gestation to birth
  Presence of IgG in umbilical cord

SECONDARY OUTCOMES:
Increase risk of neonatal morbidity | up to 30 days of life
  Respiratory distress, hypothermia, poor feeding and others
Increase risk of obstetric complications | Up to 14 days of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano, Buenos Aires, Argentina

REFERENCES:
- [Derived] Larcade R, DeShea L, Lang GA, Caballero MT, Ferretti A, Beasley WH, Tipple TE, Vain N, Prudent L, Lang ML, Polack FP, Ofman G. Maternal-Fetal Immunologic Response to SARS-CoV-2 Infection in a Symptomatic Vulnerable Population: A Prospective Cohort. J Infect Dis. 2022 Mar 2;225(5):800-809. doi: 10.1093/infdis/jiab591. PMID 34865064